CLINICAL TRIAL: NCT01308047
Title: Comparative Study of Non-inferiority Between Heavy Levobupivacaine With Enantiomeric Excess of 50% (Bupivacaine S75: R25) and Heavy Racemic Bupivacaine (Bupivacaine S50: R50) in Spinal Anesthesia for Orthopedic Procedures in the Lower Limbs.
Brief Title: Comparing Heavy Levobupivacaine With Enantiomeric Excess of 50% and Heavy Racemic Bupivacaine.
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The Sponsor has no interest in continuing the study.
Sponsor: Cristália Produtos Químicos Farmacêuticos Ltda. (Industry)
Collaborators: Irmandade da Santa Casa de Misericordia de Sao Paulo (Other); Serviço Social da Indústria do Papel, Papelão e Cortiça do Estado de São Paulo (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: CRIST016
Record Dates: First submitted 2011-02-23; First posted 2011-03-03 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Fracture of Lower Limb
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- bupivacaine S75:R25 (Experimental): 3 ml for subarachnoid block
  Interventions: Drug: Bupivacaine
- bupivacaine (S50:R50) (Active Comparator): 3 ml subarachnoid block
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Bupivacaine — single dose of 15mg by a slow injection rate of 1 ml/s
  Other Names: marcaine

SUMMARY:
The purpose of this study is to compare the non-inferiority between Heavy Levobupivacaine with Enantiomeric Excess of 50% and Heavy Racemic Bupivacaine During Spinal Anesthesia for Orthopedic Procedures in the Lower Limbs.

DETAILED DESCRIPTION:
The Heavy Levobupivacaine with Enantiomeric Excess of 50% was developed to be a safe local anesthetic replacing the Heavy Racemic Bupivacaine.

This study will evaluate the non-inferiority regarding efficacy and safety of spinal anesthesia in orthopedic procedures.

ELIGIBILITY:
Inclusion Criteria:

* ASA (American Society of Anesthesiologists) I or ASA II
* Spinal Anaesthesia for lower limb surgery
* Patient Consent

Exclusion Criteria:

* relative or absolute contraindications for spinal anesthesia
* history of hypersensitivity to the local anesthetics or components
* opioids for anesthetic adjuvant
* spinal lesions, peripheral neuropathies or any other neurologic disorders that leads to changes of sensitivity
* Body mass index = or > 35
* lumbar puncture difficulty
* ventricular extrasystoles
* dementia, others loss of cognitive ability
* difficulty in the spine
* spinal cord surgery
* anaphylactic reactions or Stevens-johnson Syndrome
* polytraumatism
* alcoholism abuse and use of illicit substance
* Changes in the blood test
* Others conditions judged by investigator's opinion

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Time of latency for sensory block at T10 dermatome. | +/- 40 min after injection
  Evaluate the sensory block at T10 after the anesthetic injection through sensory stimulation by needle.

SECONDARY OUTCOMES:
Sensory block duration | +/- 3 hours
  Verifying the duration of anesthesia from after puncture till the presence of positive sensitivity by needle stimulation region of the foot.
Motor Block Evaluation | +/- 30 min
  Motor block evaluation by Bromage Scale every five minutes after puncture till 20 minutes.
Maximum cranial dispersion verifying the largest metamer achieved. | +/- 45 min
  Evaluated by needle stimulation every 2 minutes from the removal of post-puncture needle until the maximum extension time.
Evaluation of the cardiocirculatory and respiratory parameters | +/- 8 hours
  Systolic and diastolic blood pressure (SBP and DBP), heart rate (HR), and oxygen saturation (SpO2) are evaluate during the study to measure the safety of cardiocirculatory and respiratory parameters
Time of regression of motor block by Bromage Scale | +/- 9 - 10 hours
  Will be measure the time of recovery of the motor block, the patient have to score note 4 of the Bromage Scale
The residual analgesic effect | +/- 9-10 hours
  Will be evaluated the end of the analgesic effect of the anesthetic solution when the patient asks for pain medication.
Anesthetic failure | +/- 45 min
  Evaluation of the anesthetic failure (if occur)
Adverse Events | +/- 8 - 12 hours
  During the study will be evaluate the presence of adverse event due to the anesthetic.

CONTACTS AND LOCATIONS:
Overall Officials: Ligia Mathias, PhD, Principal Investigator — Irmandade da Santa Casa de Misericórdia de São Paulo
Locations (2):
- Brazil (2):
  - Hospital Sepaco, São Paulo, São Paulo
  - Irmandade da Santa Casa de Misericórdia de São Paulo, São Paulo, São Paulo